CLINICAL TRIAL: NCT03031860
Title: Impact of Semi-quantitative Cough Strength Score as a Strong Predictor for Extubation Outcome in Head Trauma Patients: a Prospective Descriptive Study
Brief Title: Semi-quantitative Cough Strength Score (SCSS)
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor of anesthesia and ICU, Assiut University
Other Study IDs: IRB0000871237
Record Dates: First submitted 2017-01-21; First posted 2017-01-26 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semiquantitative Cough Strength Score — Evaluate extubation outcome according to degree of evaluated Semiquantitative Cough Strength Score
  Other Names: (SCSS)

SUMMARY:
Cough strength score will give true prediction of Extubation outcome

DETAILED DESCRIPTION:
Head trauma patients were evaluated for readiness to be weaned off mechanical ventilation. If they had completed an Spontaneous Breathing Trial (SBT) before extubation. To measure Semiquantitative Cough Strength Score (SCSS), the investigator will put the patients at 30° to 45°, measure SCSS, first. The investigator enhance the patient to cough with as much effort as, when the investigator disconnect the ventilator. The cough strength was scored from 0 to 5 as follows: 0 = no cough on command, 1 = audible movement of air through the endotracheal tube but no audible cough, 2 = weakly (barely) audible cough, 3 = clearly audible cough, 4 = stronger cough and 5 = multiple sequential strong coughs.

ELIGIBILITY:
Inclusion Criteria:

* The study included 80 adult male and female patients' their ages between 18-65 years admitted to trauma ICU with head trauma, on mechanical ventilation more than 24 hours and was ready to be weaned off from mechanical ventilation after successful spontaneous breathing trial and Glasgow Coma Scale (GCS) score > 8 before extubation

Exclusion Criteria:

• Patients who had undergone tracheostomy before extubation, GCS ≤ 8, chest trauma (ribs fracture and lung contusion) and patients with chronic chest disease (Chronic obstructive pulmonary disease, tuberculosis and cancer lung) were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample of this study include 80 head trauma patients from both sex of critically ill mechanically ventilated patient admitted to trauma Intensive Care Unit (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Extubation outcome (success or failure), is the patient reintubate again or not and it's correlation with the level of Cough Strength Score | within 6 hours postextubation
  The cough strength was scored from 0 to 5 as follows: 0 = no cough on command, 1 = audible movement of air through the endotracheal tube but no audible cough, 2 = weakly (barely) audible cough, 3 = clearly audible cough, 4 = stronger cough and 5 = multiple sequential strong coughs.

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Aziz, Principal Investigator — assiut university faculty of nursing
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White AC. Long-term mechanical ventilation: management strategies. Respir Care. 2012 Jun;57(6):889-97; discussion 898-9. doi: 10.4187/respcare.01850. PMID 22663965